CLINICAL TRIAL: NCT04070053
Title: Treatment of Hypoxemic Respiratory Failure and ARDS With Protection, Paralysis, and Proning (TheraPPP) Pathway: a Pilot Before and After Study
Brief Title: Treatment of Hypoxemic Respiratory Failure and ARDS With Protection, Paralysis, and Proning (TheraPPP) Pathway
Acronym: TheraPPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Ken Kuljit Parhar, MD, Consultant Intensivist & Clinical Assistant Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB19-0939; 897 (Other Grant/Funding Number: M.S.I. Foundation); 2019 (Other Grant/Funding Number: Chief Medical Office (CMO) Alberta Health Services)
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Acute Respiratory Distress Syndrome; Hypoxemic Respiratory Failure; ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: We will perform a before and after study to evaluate the feasibility and acceptability of the HRF and ARDS Pathway during its pilot implementation. All mechanically ventilated patients will enter the pathway during the one month implementation period and one year post-implementation period.
  To assess Pathway feasibility we will collect patient data for two years and one month: one year immediately prior to implementation as well as one month during plus one year following implementation.
  To assess acceptability of the pathway we will conduct a survey to clinicians who used the pathway.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TheraPPP Pathway (Experimental): We will perform a before and after study to evaluate the feasibility and acceptability of the HRF and ARDS Pathway during its pilot implementation.
  All mechanically ventilated patients will enter the pathway during the one month implementation and one year post-implementation periods.
  To assess Pathway feasibility we will collect patient data for approximately two years and one month: one year immediately prior to implementation, one month during, and one year following implementation.
  To assess acceptability of the pathway we will conduct a survey to clinicians who used the Pathway.
  Interventions: Other: TheraPPP Pathway

INTERVENTIONS:
Other: TheraPPP Pathway — TheraPPP Steps:
  Step 1. All mechanically ventilated patients will have a height measured and documented. Step 2. Screening for HRF. Step 3. Initiate Lung Protective Ventilation (LPV). Step 4. Paralysis. Step 5. Prone Positioning.

SUMMARY:
Treatment of patients with Hypoxemic respiratory failure (HRF) and Acute Respiratory Distress Syndrome (ARDS) is complex. Therapies that have been shown to save the lives of patients with HRF and ARDS are available but they are not always provided. To reduce practice variation and improve adherence to evidence-informed therapies, the investigators developed the Treatment of Hypoxemic Respiratory Failure (HRF) and ARDS with Protection, Paralysis, and Proning (TheraPPP) Pathway.

The purpose of this pilot study is to test the feasibility and acceptability of the TheraPPP Pathway. To assess feasibility, the investigators will test the ability to measure adherence to the pathway as well as patient and economic outcomes. To assess perceptions about the acceptability of the TheraPPP Pathway, the investigators will conduct a survey to clinicians who used the Pathway.

DETAILED DESCRIPTION:
Hypoxemic respiratory failure (HRF) and ARDS are common conditions among patients admitted to the Intensive care unit (ICU). Treatment of these patients is complex. Evidence based therapies that can improve survival exist; however, implementation is extremely inconsistent. As a potential solution to this problem, the investigators developed the Treatment of Hypoxemic Respiratory Failure (HRF) and ARDS with Protection, Paralysis, and Proning (TheraPPP) Pathway to reduce practice variation and improve adherence to evidence-informed therapy. The objective of this pilot before and after study is to evaluate the feasibility and acceptability of the TheraPPP Pathway.

The pilot study will use a before and after quasi-experimental design to evaluate the feasibility and acceptability of the TheraPPP pathway. The TheraPPP pathway is a comprehensive evidence-based, stakeholder-informed pathway for the diagnosis and management of HRF. The study will be conducted in a single center mixed medical surgical ICU. The study population will include all patients who are admitted to the ICU and are mechanically ventilated.

The pathway will be implemented over a one month period, followed by a one year post implementation assessment period. The comparison (control) therapy will be usual management assessed in the one year pre-implementation period. We estimate approximately 1000 patients will be included in the study.

The primary objectives of the pilot study will be to assess feasibility and acceptability. To assess feasibility, the investigators will test the ability to measure: (1) Fidelity through 5 process of care indicators (2) Patient and economic outcomes. To assess the acceptability of the Pathway, the investigators will conduct a survey to clinicians who used the pathway. The acceptability survey will be sent to approximately 250 ICU clinicians.

For data analysis, no specific comparisons will be made as the investigators are testing the ability to measure the outcomes. However, feasibility and acceptability data will be presented in aggregate as frequency with proportion or median with interquartile range, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Foothills Medical Center Intensive Care Unit (Pod A)
* Invasively mechanically ventilated

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
FEASIBILITY (Fidelity) Fidelity of the intervention using a composite fidelity score | 4 months (after the post-implementation period)
  The composite fidelity score is measured daily for each patient. It is scored out of 5 and awards 1 point for each fidelity indicator (listed below) that investigators are able to measure,
  1. If ventilated ≥24 hours, is a height measured (step 1)
  2. If arterial to inspired oxygen ratio (PaO2:FiO2 ratio or PF ratio) ≤300, is the medial tidal volume ≤8mL/kg stratified by volume and pressure control (step2/3)
  3. If PF ratio ≤300, is a plateau pressure measured (step 3)
  4. IF patient has HRF and PF ratio ≤150, was neuromuscular blockade used in that 24 hour period (step 4)
  5. If the patient has HRF and PF ratio ≤150 and FiO2 ≥0.6, did the patient receive prone ventilation (step 5).
FEASIBILITY (Economic) Cost per safe ventilation day | 4 months (after the post-implementation period)
  Cost per safe ventilation day from the perspective of the health care system
ACCEPTABILITY Pathway Acceptability measured using the Theoretical Framework of Acceptability (TFA) | 4 months (after the post-implementation period)
  The primary outcome for acceptability is the proportion of seven TFA constructs (7 constructs of acceptability) graded with a median score of 5 or above from a 7-point Likert scale, indicating agreement.

SECONDARY OUTCOMES:
The proportion of ventilated patients with a height measured | 4 months (after the post-implementation period)
  Total number of ventilated patients with a height measured divided by the total number of ventilated patients
The proportion of ventilated patients with a height measured within 1 hour of admission | 4 months (after the post-implementation period)
  Total number of ventilated patients with a height measured within 1 hour of admission divided by the total number of ventilated patients
The proportion of patients ventilated ≥24 hours with a height measured | 4 months (after the post-implementation period)
  Total number of ventilated patients for ≥24 hours with a height measured divided by the total number of ventilated patients ≥24 hours
The median time to height measurement from admission | 4 months (after the post-implementation period)
  The median time to height measurement from admission for patients ventilated ≥24 hours
The proportion of patient days with arterial to inspired oxygen ratio(PaO2:FiO2 ratio or PF ratio) ≤300 with a tidal volume ≤8mL/kg stratified by volume and pressure control | 4 months (after the post-implementation period)
  The total number of patient days with arterial to inspired oxygen ratio(PaO2:FiO2 ratio or PF ratio) ≤300 with a tidal volume ≤8 mL/kg divided by the total number of of patient days with arterial to inspired oxygen ratio(PaO2:FiO2 ratio or PF ratio) ≤300 stratified by volume and pressure control
The proportion of patient days with PF ratio ≤300 with a plateau pressure measured | 4 months (after the post-implementation period)
  The total number of patient days with PF ratio ≤300 with a plateau pressure measured divided by the total number of patient days with PF ratio ≤300
The proportion of patient days with HRF and PF ratio ≤150 who receive neuromuscular blockade | 4 months (after the post-implementation period)
  The number of patient days with HRF and PF ratio ≤150 who receive neuromuscular blockade divided by the number of patient days with HRF and PF ratio ≤150
The proportion of patient days with HRF and PF ratio ≤100 who receive neuromuscular blockade | 4 months (after the post-implementation period)
  The number of patient days with HRF and PF ratio ≤100 who receive neuromuscular blockade divided by the number of patient days with HRF and PF ratio ≤100
The proportion of patient days with HRF and PF ratio ≤150 and FiO2 ≥0.6 receiving prone ventilation | 4 months (after the post-implementation period)
  The number of patient days with HRF and PF ratio ≤150 and FiO2 ≥0.6 receiving prone ventilation divided by the number of patient days with HRF and PF ratio ≤150 and FiO2 ≥0.6
The proportion of patient days with HRF and PF ratio ≤100 and FiO2 ≥0.6 receiving prone ventilation | 4 months (after the post-implementation period)
  The number of patient days with HRF and PF ratio ≤100 and FiO2 ≥0.6 receiving prone ventilation divided by the number of patient days with HRF and PF ratio ≤100 and FiO2 ≥0.6
Days of safe ventilation for females | 4 months (after the post-implementation period)
  Days of safe ventilation for females (proportion of days of safe ventilation with a median daily tidal volume ≤ 8 mL/kg predicted body weight)
Number of patients who do not survive | 4 months (after the post-implementation period)
  Number of patients who die in the ICU, hospital, and at or before 28-day hospital
Number of ventilator-free days (VFDs) 28-day ventilator-free days (VFDs) | 4 months (after the post-implementation period)
  Number of days that patients are not on the ventilator
The proportion of patients receiving rescue therapies | 4 months (after the post-implementation period)
  The proportion of patients receiving rescue therapies including inhaled vasodilators, Extracorporeal Life Support.
Total cost for the ICU admission | 4 months (after the post-implementation period)
  Total cost for the ICU admission
Total cost for the index hospitalization | 4 months (after the post-implementation period)
  Total cost for the index hospitalization
Length of Stay (LOS) (ICU, hospital) / the number of days that patients stay in the ICU and in hospital | 4 months (after the post-implementation period)
  The number of days that patients stay in the ICU and in hospital
Days of safe ventilation | 4 months (after the post-implementation period)
  Days of safe ventilation (proportion of days of safe ventilation with a median daily tidal volume ≤ 8 mL/kg predicted body weight)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Parhar, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Hospital Intensive Care Unit, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No